CLINICAL TRIAL: NCT06696638
Title: Physiological Effects of Lung Impedance Tomography-guided and Plat Pressure-guided Phigh During Airway Pressure Release Ventilation in Patients With Acute Respiratory Distress Syndrome
Brief Title: Physiological Effects of Lung Impedance Tomography-Guided and Plat Pressure-Guided Phigh During APRV in Patients With ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XiaoJing Zou,MD (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, XiaoJing Zou,MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: APRVPhigh2024
Record Dates: First submitted 2024-11-13; First posted 2024-11-20 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: ARDS: Acute Respiratory Distress Syndrome
Keywords: ARDS; APRV; EIT; Phigh
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention group (Experimental): EIT-guided Phigh settings during APRV
  Interventions: Device: EIT-guided Phigh settings during APRV
- Control group (No Intervention): Pplat-guided Phigh settings during APRV

INTERVENTIONS:
Device: EIT-guided Phigh settings during APRV — The Phigh level selected for the patients in the Intervention group was the intercept point of cumulated collapse and overdistension percentage curves, providing the best compromise between collapsed and overdistended lung.
  Arms: Intervention group

SUMMARY:
This study aims to investigate the effects of EIT-guided and Pplat-guided Phigh settings on regional ventilation and perfusion in ARDS patients during APRV, while also examining the impact of different Phigh settings on gas exchange, respiratory mechanics, and hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ARDS according to the 2023 global new definition of ARDS.
* Age ≥ 18 years.

Exclusion Criteria:

* Severe chronic obstructive pulmonary disease, severe asthma, pulmonary bullae, pneumothorax, subcutaneous emphysema, mediastinal emphysema, etc. · Contraindications for EIT, such as chest wound dressing, pacemaker implantation, defibrillator use, etc.
* Pulmonary interstitial disease.
* Uncorrected shock of various types.
* Intracranial hypertension.
* Pregnant and postpartum women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The effects of Phigh guided by different methods on regional lung ventilation assessed by EIT | 1 Hour Post-Intervention

SECONDARY OUTCOMES:
Global inhomogeneity assessed by electrical impedance tomography | 1 Hour Post-Intervention
Center of ventilation assessed by electrical impedance tomography | 1 Hour Post-Intervention
ventilation/perfusion matching assessed by EIT | 1 Hour Post-Intervention
Respiratory system compliance | 1 Hour Post-Intervention
  Tidal volume divided by plateau pressure
mean arterial pressure | 1 Hour Post-Intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No